CLINICAL TRIAL: NCT01805128
Title: EXPLORATION OF THE SOCIAL COGNITION IN ADOLESCENTS WITH A Dissociative Disorder OR AUTISM SPECTRUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Centre Hospitalier d'Antibes Juans les Pins (Unknown); Centre Hospitalier de Cannes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 12-AOI-04
Record Dates: First submitted 2013-02-22; First posted 2013-03-06 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Schizophrenia; Autistic Disorder
Keywords: Schizophrenia; Autistic Disorder; social cognition
MeSH Terms: conditions — Schizophrenia; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- schizophrenia (Experimental): child with a DSM-IV diagnosis of schizophrenia
  Interventions: Other: Facial recognition of emotions; Other: understanding metaphors; Other: Attribution of intentionality to others in social situations depending on the type of situation
- autism spectrum disorder (Experimental): child with a DSM-IV diagnosis of autism spectrum disorder
  Interventions: Other: Facial recognition of emotions; Other: understanding metaphors; Other: Attribution of intentionality to others in social situations depending on the type of situation
- Healthy (Experimental): child having no DSM-IV diagnosis of schizophrenia spectrum disorder or autism
  Interventions: Other: Facial recognition of emotions; Other: understanding metaphors; Other: Attribution of intentionality to others in social situations depending on the type of situation

INTERVENTIONS:
Other: Facial recognition of emotions — The purpose is to consider the recognition of emotions expressed on face in patients with a schizophrenic disorder, autism and in healthy subjects.
Other: understanding metaphors — Explore understanding of figurative language, including metaphor, in schizophrenic patients, autistic and healthy, and well understand how patients develop an interpretation from access to speaker's communicative intentionality (theory mind).
Other: Attribution of intentionality to others in social situations depending on the type of situation — Compare the style of attribution of intentions in three populations of subjects: schizophrenic, autistic and healthy.

SUMMARY:
The schizophrenic disorders and pervasive developmental disorders are neurodevelopmental disorders distinct origin who share common challenges to engage and maintain social relationships and mutual disturbances of affective contact. An important issue of research is to determine the cognitive and brain mechanisms underlying social disability in these two pathologies. Several lines of social cognition have been systematically explored: the perception of emotions, the ability to attribute intentionality and mental states to others (theory of mind), the understanding of social situations in different contexts. We made the observation today that research findings clearly in the field of autism and schizophrenic disorders that converge on common patterns neurocognitive abnormalities. Consequently, many programs support published today use the same therapeutic targets and the same tools in both pathologies. This raises two questions of science: (1) whether the disorders of social cognition reported in the field of autism and schizophrenia are "specific deficit" and not "specific condition", that is to say they are inherent social disadvantage whatever condition or (2) if these disorders of social cognition is a pattern common to autism and schizophrenia but are the result of specific neurocognitive mechanisms and different in each these pathologies. Systematic exploration of these issues is a current issue for understanding the pathophysiological borders between the two neurodevelopmental disorders but also to better define the potential targets of therapeutic strategies, psycho-educational and remediation of disorders of social cognition in autism and schizophrenia.

Main objective: To compare clinical cognitive profiles in adolescents with a schizophrenic disorder, autistic or healthy in the three areas of social cognition: perception of emotions, attribution of intentions to others (theory of mind) and style attribution. We shall constitute three population groups of patients, a group of patients meeting the diagnosis of schizophrenia, a group of patients with autism and a control group (healthy subjects).

DETAILED DESCRIPTION:
The schizophrenic disorders and pervasive developmental disorders are neurodevelopmental disorders distinct origin who share common challenges to engage and maintain social relationships and mutual disturbances of affective contact. An important issue of research is to determine the cognitive and brain mechanisms underlying social disability in these two pathologies. Several lines of social cognition have been systematically explored: the perception of emotions, the ability to attribute intentionality and mental states to others (theory of mind), the understanding of social situations in different contexts. We made the observation today that research findings clearly in the field of autism and schizophrenic disorders that converge on common patterns neurocognitive abnormalities. Consequently, many programs support published today use the same therapeutic targets and the same tools in both pathologies. This raises two questions of science: (1) whether the disorders of social cognition reported in the field of autism and schizophrenia are "specific deficit" and not "specific condition", that is to say they are inherent social disadvantage whatever condition or (2) if these disorders of social cognition is a pattern common to autism and schizophrenia but are the result of specific neurocognitive mechanisms and different in each these pathologies. Systematic exploration of these issues is a current issue for understanding the pathophysiological borders between the two neurodevelopmental disorders but also to better define the potential targets of therapeutic strategies, psycho-educational and remediation of disorders of social cognition in autism and schizophrenia.

Main objective: To compare clinical cognitive profiles in adolescents with a schizophrenic disorder, autistic or healthy in the three areas of social cognition: perception of emotions, attribution of intentions to others (theory of mind) and style attribution. We shall constitute three population groups of patients, a group of patients meeting the diagnosis of schizophrenia, a group of patients with autism and a control group (healthy subjects).

Inclusion criteria: patients aged 12 to 18, with a verbal IQ greater than or equal to 70, a DSM-IV diagnosis of autism and / or schizophrenia.

Assessment instruments: (1) clinical assessment instruments using standardized structured interviews that have already shown good sensitivity in our preliminary studies (2) techniques neuro-social cognition scientifically validated by the expert group of the ANR we are partners.

The study of active files and preliminary results, we can estimate the population to 20 patients per group, a total of 60 patients.

The originality of this study focuses on the ability to compare two populations in the same field of social cognition in three dimensions, which hitherto have been explored separately in the literature. The expected results are a range of prevention and treatment of major psychiatric children and adolescents because they help define therapeutic targets specific to each population

ELIGIBILITY:
Inclusion Criteria:

* Child with a DSM-IV diagnosis of schizophrenia or autism spectrum disorder:

  * Schizophrenic patients, positive to the award of psychosis section of the Kiddie SADS and having a negative ADI.

or:

* Patients with autism spectrum disorder, diagnosed by the scale ADI (Autism Diagnostic Interview) or ADOS (Autism Diagnostic Observation Schedule): Autism Asperger and PDD nos. These patients do not respond to a diagnosis of psychosis Kiddie-SADS according.

  * Total IQ greater than or equal to 70

Exclusion Criteria:

* Genetic disorders, neurological and neurosensory
* Child satisfy both the diagnosis of autism spectrum disorder and schizophrenia than (comorbidity).
* Will not be included patients who participate in a study on rehabilitation for social skills.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Compare cognitive profiles in clinical adolescents with a schizophrenic disorder, autistic or healthy in the three areas of social cognition | First day
  Compare cognitive profiles in clinical adolescents with a schizophrenic disorder, autistic or healthy in the three areas of social cognition: the perception of emotions, attribution of intentions to others (theory of mind) and style attribution.
  We will study the brain evoked potentials during the execution of the task of facial emotion recognition.

SECONDARY OUTCOMES:
Compare the cognitive profiles within the clinical group of schizophrenic | First day
  Compare the cognitive profiles within the clinical group of schizophrenic patients, depending on the type of schizophrenia presented (as positive, negative or disorganized).
  For the study of attribution of intentions to others: This is to test the understanding of metaphors patients. Three types of statements are presented: forward literals, metaphorical statements and statements incongruous; patients should judge the plausibility semantics of these sentences. We study the behavioral and electrophysiological data.
Cognitive profiles compare clinical results between the different types of schizophrenia and autism patients. | First day
  Cognitive profiles compare clinical results between the different types of schizophrenia and autism patients.
  Self-assessment in the form of a questionnaire with several social situations of everyday life. The subject must plan and assign intentionality to a character. We get scores dimensions studied.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle DOR, Medical Doctor, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (3):
- France (3):
  - Centre Hospitalier d'Antibes Juans les Pins, Antibes
  - Centre hospitalier de Cannes, Cannes
  - CHU de Nice, Nice